CLINICAL TRIAL: NCT06433713
Title: Effect of Intraoperative Intravenous Lidocaine on Postoperative Pain and Return of Bowel Function After Cesarean Sections, a Double-blinded Randomized Control Study
Brief Title: Effect of Intraoperative Intravenous Lidocaine on Postoperative Pain and Return of Bowel Function After Cesarean Sections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Fathy Zaky, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-220
Record Dates: First submitted 2024-04-24; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Postoperative Return of Bowel Function
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine Group (Experimental): Intravenous lidocaine infusion, 2 mg/kg/hour
  Interventions: Drug: Lidocaine IV
- Control Group (Placebo Comparator): Normal saline infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine IV — They received IV infusion of 2 mg/kg per hour of lidocaine starting with skin incision, which was maintained until skin closure. This was done using a syringe pump with the calculated amount of lidocaine added to 50 ml of normal saline infused at a rate of 50 ml/hr.
  Arms: Lidocaine Group
Drug: Placebo — 0.9% normal saline infusion
  Other Names: Normal saline
  Arms: Control Group

SUMMARY:
Postoperative discomfort is a frequently seen adverse event after to caesarean operation. Early mobilization and bonding of the mother and her infant are typically impacted by this phenomenon.

Nevertheless, the current state of postoperative analgesia and recovery remains inadequate in clinical settings. In the context of major abdominal surgery, opioids are often regarded as the preferred postoperative analgesic. Nevertheless, they possess adverse side effects that might impact the process of recuperation after surgery. These symptoms include nausea and vomiting, decreased bowel movement, and shallow breathing.

One additional challenging consequence after surgery is the delayed restoration of bowel function, which has the potential to extend the duration of hospitalization and impede the initiation of oral feeding, resulting in gaseous colonic distension.

The administration of lidocaine infusion has been shown to possess analgesic, anti-hyperalgesic, and anti-inflammatory characteristics.

The use of intravenous lidocaine after surgery is postulated to have the dual effect of mitigating postoperative pain and expediting the resumption of bowel movements.

Recent studies have shown that the administration of intravenous lidocaine, either as a single dosage or by continuous infusion, may have potential advantages in maintaining gastrointestinal motility and exerting an impact on biochemical pain mechanisms.

However, the literature presents contradictory data about the effectiveness of lidocaine in providing sufficient postoperative pain relief and reducing postoperative ileus.

Consequently, this study was conducted and aimed to assess the effect of intravenous intraoperative lidocaine on postoperative pain and early return of bowel function following elective caesarean section.

This randomized clinical trial was conducted at Obstetrics and Gynecology Department, Faculty of Medicine, Cairo University Hospitals from August till December 2023. A total of 60 pregnant women underwent elective caesarean section were enrolled and randomized into two groups; experimental group who received IV infusion of lidocaine starting with skin incision, which was maintained until skin closure and control group who received 0.9% normal saline at the same rate as that described in the experimental group. Both groups were compared as regard total operative time, medications given, start-stop time of the study drug infusion, and degree of pain using visual analogue scale, need for analgesics, time for first healing of normal intestinal sounds and time to first flatus and symptoms of lidocaine toxicity were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. American society of anesthesiology (ASA) class II (Normal pregnancy, well controlled gestational HTN, controlled preeclampsia without severe features, diet-controlled gestational DM).
3. Singleton term pregnancy.
4. Elective caesarean section.
5. Spinal anesthesia.

Exclusion Criteria:

1. Atypical postoperative care e.g. following caesarean hysterectomy.
2. Inflammatory bowel disease.
3. Prolonged surgery >1.5 hours.
4. Medical disorders e.g. liver or renal affection
5. Previous bowel surgery.
6. History' of allergic reaction to lidocaine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Effect of intraoperative intravenous lidocaine on visual analogue scale pain scores among the two groups. | 12-24 hours
  The patients are asked to describe how much pain they feel in a scale from 0 to 10. Minimum score 0, maximum score 10 where 10 is worse and means more pain
Effect of intraoperative intravenous lidocaine on early return of bowel function assessed by the time to first hearing of bowel sounds and the time to first flatus passing. | 12-24 hours
  Time to hearing of bowel sounds, passing of flatus & passing of stool

SECONDARY OUTCOMES:
Occurrence of lidocaine toxicity with the standard dose given. | 12-24 hours
  Nausea, perioral numbness, neurological symptoms or cardiac arrhythmia
Duration of hospital stay. | 12-24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Kasr Al Aini School of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided